CLINICAL TRIAL: NCT01849965
Title: A Randomized, Double-Blind, Parallel-group, Vehicle and Standard of Care-controlled Phase 3 Clinical Trial to Evaluate the Efficacy and Safety of DSC127 in Treating Non-healing Foot Ulcers in Subjects With Diabetes Mellitus
Brief Title: Phase 3 Study Evaluating Efficacy and Safety of DSC127 Compared With Vehicle and With Standard-of-care in Diabetic Foot Ulcers
Acronym: STRIDE 2
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Integra LifeSciences Corporation (Industry)
Collaborators: Integrium (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DSC127-2012-02
Record Dates: First submitted 2013-05-06; First posted 2013-05-09 (Estimated); Last update posted 2017-12-12 (Actual); Status verified 2017-12

CONDITIONS: Diabetic Foot Ulcers
Keywords: diabetic foot ulcers; Wagner Grade 1 or 2 ulcers
MeSH Terms: conditions — Diabetic Foot | interventions — aclerastide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- DSC127 (Active Comparator): DSC127 0.03% in a vehicle gel (hydroxyethyl cellulose (HEC) with parabens)
  Interventions: Drug: DSC127
- Vehicle gel (Placebo Comparator): Vehicle gel comprising HEC with parabens
  Interventions: Drug: placebo vehicle gel
- Standard of Care gel (Placebo Comparator): Aquasite gel, as standard of care gel
  Interventions: Drug: Standard of Care gel, Aquasite

INTERVENTIONS:
Drug: DSC127 — DSC127 0.03%, daily topical application to diabetic foot ulcer for a period of up to 28 days or until ulcer closure, whichever occurs sooner.
  Arms: DSC127
Drug: placebo vehicle gel
  Arms: Vehicle gel
Drug: Standard of Care gel, Aquasite
  Arms: Standard of Care gel

SUMMARY:
To determine if aclerastide (DSC127) is effective in increasing incidence of complete wound closure up to 10 weeks confirmed 2 weeks later, compared with vehicle (gel without active ingredient) and compared with a standard-of-care gel, in subjects with diabetes mellitus (DM) who have chronic Wagner Grade 1 or 2 diabetic foot ulcers, 0.75 - 6cm2 in size.

DETAILED DESCRIPTION:
Subjects will undergo a two week screening period to assess plantar ulcer healing, and those healing less than 30% will be eligible for randomization providing all other criteria are met. Four weeks of "blinded" randomized treatment follows the screening period, and an observation period of six weeks follows the treatment period. If the ulcer closes during the treatment or observation period, the closure will be confirmed at a visit two weeks later, and at this time the subjects enters a durability assessment period of up to 12 weeks.

All aspects of Standard of Care are followed throughout the study period.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ambulatory subject age ≥18 years at the time of informed consent
* Has type 1 or type 2 DM under metabolic control as confirmed by a glycosylated hemoglobin (HbA1c) of ≤12% and a serum creatinine level of ≤3mg/dL
* At Screening and Baseline (prior to randomization), subject has at least one ulcer that fulfills all of the following criteria:

  * present for ≥1 month and ≤1 year
  * Partial- or full- thickness and not involving bone, tendon, or capsule (probing to tendon or capsule), i.e. Wagner Grade 1 or 2.
  * Has no sign of infection or osteomyelitis
  * Plantar neuropathic ulcer - predominately be on the plantar surface (i.e. weight bearing) of the foot to ensure adequate off-loading and may include the toes
  * Size of the target ulcer must be 0.75-6 cm2.
  * Target ulcer must be non-healing as defined as <30% reduction in area in response to standard of care during the Screening Period

    * If more than one ulcer is present that meets the inclusion criteria, the largest one will be considered the target ulcer
    * If there are two ulcers of the same size that meet all criteria, the one with the higher Wagner Grade will be considered the target ulcer
    * If there are two ulcers of the same size and the same Wagner Grade, the one present for the longest qualifying time will be the target ulcer.
    * Non-target ulcers will also be treated according to standard of care (Acute Charcot Neuroarthropathy of the foot with the target ulcer must be excluded)
* Has an ankle brachial index (ABI) ≥0.7 on the foot with the target ulcer.
* Has an assessment of the baseline level of neuropathy of the foot using Semmes-Weinstein filaments.
* A female subject of childbearing potential must have a negative serum pregnancy test at the time of Screening.
* A female subject of childbearing potential must be willing to use a medically acceptable method of birth control, such as Essure®, hormonal contraception (oral pills, implantable device, or skin patch), intrauterine device, tubal ligation, or double barrier throughout the study. A female subject of childbearing potential who practices abstinence is not required to employ birth control.
* Has the ability and willingness to understand and comply with study procedures and to give written informed consent prior to enrollment in the study or initiation of study procedures

Exclusion Criteria:

* Has a known hypersensitivity to any of the investigational drug or vehicle or standard of care gel components
* Has been exposed to any investigational agent within 30 days of entry into the study
* A female who is pregnant or nursing
* Has active malignant disease of any kind except for basal cell carcinoma (of the skin). A subject, who has had a malignant disease in the past, was treated and is currently disease-free, may be considered for study entry.
* Has a hemoglobin of less than 8.5 gm/dL.
* Transaminase levels greater than 3 × normal
* Is receiving hemodialysis or chronic ambulatory peritoneal dialysis (CAPD) therapy
* Has had prior radiation therapy to any part of the foot with the target ulcer under study
* Use of systemic corticosteroids and immunosuppressants (within the 8 weeks prior to screening)
* Has an ulcer primarily ischemic in etiology
* Has sickle-cell anemia, Reynaud's, or peripheral vascular disease
* Has received a biologic agent, growth factor, or skin equivalents (Regranex®, Apligraft, or Dermagraft), in the past 30 days
* Has a target ulcer which is determined to be clinically infected and requires antimicrobials. Any antibiotic therapy must be completed or discontinued at Screening.
* Has a Wagner Grade 3 or higher DFU, deep abscess, or gangrene
* Has uncontrolled hypertension, in the opinion of the Investigator.
* Any other finding, which in the opinion of the Investigator, may interfere with the assessment of the product or participation of the patient in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 396 (Actual)
Dates: Start 2013-04; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
The proportion of subjects with a target ulcer which achieves complete wound closure by 10 weeks (confirmed 2 weeks later) after initiation of treatment. | Target ulcer must achieve complete wound closure by 10 weeks post first treatment
  Primary endpoint of complete closure is assessed by the Principal Investigator at the site; ulcer measurements are calculated via tracings submitted to the Canfield system, and photographs are collected as confirmation of closure via the Canfield system. Assessment of aclerastide (DSC127) vs vehicle control.

SECONDARY OUTCOMES:
The proportion of subjects with a target ulcer which achieves complete wound closure by 10 weeks (confirmed two weeks later) after initiation of treatment. | Target ulcer must achieve complete wound closure by 10 weeks post first treatment
  Primary endpoint of complete closure is assessed by the Principle Investigator at the site; ulcer measurements are calculated via tracings submitted to the Canfield system, and photographs are collected as confirmation of closure via the Canfield system. Assessment of aclerastide (DSC127) vs Standard of Care control.

OTHER OUTCOMES:
Time to the visit where the target ulcer achieves confirmed complete wound closure | Measurements to ten weeks post first dose
Percent reduction in target ulcer area per week. | Up to ten weeks post first dose
Incidence of and time to target ulcer recurrence after confirmed complete wound closure has been established. | To a maximum of 24 weeks post first dose

CONTACTS AND LOCATIONS:
Overall Officials: Alan Dunton, MD, Study Director — Integra LifeSciences Corporation
Locations (56):
- United States (33):
  - East Valley Foot and Ankle Specialist, Mesa, Arizona
  - Arizona Burn Center Maricopa Medical Center, Phoenix, Arizona
  - Associated Foot & Ankle Specialists, PC, Phoenix, Arizona
  - Ledesma Foot and Ankle, Phoenix, Arizona
  - Precision Trials, Phoenix, Arizona
  - Center for Clinical Research, Inc., Castro Valley, California
  - Reliance Institute of Clinical Research, Chino, California
  - Vladimir Zeetser, DPM, Encino, California
  - Innovative Medical Technologies, LLC, Los Angeles, California
  - Samuel Merritt University, California School of Podiatric Medicine, Oakland, California
  - Center for Clinical Research, Inc., San Francisco, California
  - The Diabetic Foot and Wound Center, Denver, Colorado
  - Orthopedic Research Associates, Boynton Beach, Florida
  - Invesclinic, LLC, Fort Lauderdale, Florida
  - Research in Miami, Inc., Hialeah, Florida
  - River City Clinical Research, Jacksonville, Florida
  - Advanced Pharma CR, LLC, Miami, Florida
  - University of Miami, Miami, Florida
  - Phoenix Medical Research, Miami, Florida
  - New Phase Clincal Trials, Inc., Miami Beach, Florida
  - Bluegrass Foot Center c/o Research Concierge, LLC, Owensboro, Kentucky
  - Grace Research, Shreveport, Louisiana
  - American Center for Clinical Trials, Southfield, Michigan
  - Dr. Vincent Giacalone, Emerson, New Jersey
  - Wayne Memorial Hospital, Goldsboro, North Carolina
  - O'Malley Foot and Ankle, Wilmington, North Carolina
  - Regional Infectious Disease & Infusion Center Inc., Lima, Ohio
  - Paddington Testing Clinic, Philadelphia, Pennsylvania
  - Martin Foot & Ankle, York, Pennsylvania
  - North Texas Podiatric Medicine & Surgery, Dallas, Texas
  - Bone and Joint Institute, Fort Worth, Texas
  - Houston Foot & Ankle Specialists, Houston, Texas
  - Redwood Health Center, Salt Lake City, Utah
- Canada (5):
  - The Mayer Institute, Hamilton, Ontario
  - Lawson Health Research Institute, London, Ontario
  - Xceed Clinical, Whitby, Ontario
  - Centre Podiatrique et Soins des Plaies, Boucherville, Quebec
  - Centre de recherche du CHUS, Sherbrooke, Quebec
- Puerto Rico (4):
  - Centro de Curacion de Heridas del Caribe, Inc., Aguadilla
  - Office of Renier D. Gonzalez-Cruz, MD, Juana Díaz
  - Clinical Research Puerto Rico, San Juan
  - Wound and Ulcer Care Clinic, San Juan
- South Africa (14):
  - GCT - Mercantile Clinical Trial Centre - Primecure Clinic, Port Elizabeth, Eastern Cape
  - Iatros International, Bloemfontein, Free State
  - Josha Research, Bloemfontein, Free State
  - Worthwhile Clinical Trials, Benoni, Gauteng
  - Dr Lakha's Consulting Rooms, Johannesburg, Gauteng
  - Newtown Clincal Research Centre, Newtown, Gauteng
  - Sunninghill Hospital, Sunninghill, Gauteng
  - Synapta Clinical Research Centre, Durban, KwaZulu-Natal
  - Flamco Clinical Trials, Durban, KwaZulu-Natal
  - Brookedale Clinical Research Centre, Phoenix, KwaZulu-Natal
  - Tiervlei Trial Centre, Karl Bremer Hospital, Cape Town, Western Cape
  - Tread Research, Parow, Western Cape
  - Boland Ethical Research Group, Worcester, Western Cape
  - Randles Road Medical Centre, Durban, ZwaZulu Natal